CLINICAL TRIAL: NCT00808613
Title: Prospective, Single-center, Non-randomized, Consecutive Series Study Comparing Functional Differences Between a Standard Posterior Stabilized TKR and a High-flexion Posterior Stabilized TKR
Brief Title: Optetrak Posterior Stabilized Versus Optetrak Hi-Flex
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study withdrawn prior to initiation
Sponsor: Exactech (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR07-001
Record Dates: First submitted 2008-12-15; First posted 2008-12-16 (Estimated); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Arthropathy of Knee; Arthritis and/or Post-traumatic Degenerative Problems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Optetrak Posterior Stabilized TKR (Active Comparator): Subjects in this arm will receive an Optetrak Posterior Stabilized total knee system.
  Interventions: Device: Optetrak PS
- Optetrak Hi-Flex TKR (Active Comparator): Subjects in this arm will receive an Optetrak Hi-Flex total knee system.
  Interventions: Device: Optetrak Hi-Flex

INTERVENTIONS:
Device: Optetrak PS — Optetrak Posterior Stabilized total knee replacement
  Arms: Optetrak Posterior Stabilized TKR
Device: Optetrak Hi-Flex — Optetrak Hi-Flex total knee replacement
  Arms: Optetrak Hi-Flex TKR

SUMMARY:
The purpose of this study is to evaluate the differences in clinical outcomes between the Optetrak® Posterior Stabilized ("Optetrak® PS", Exactech, Gainesville, FL) and the Optetrak® Hi-Flex™ ("Optetrak® HF", Exactech, Gainesville, FL) knee designs.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the differences in clinical outcomes between the Optetrak® Posterior Stabilized ("Optetrak® PS", Exactech, Gainesville, FL) and the Optetrak® Hi-Flex™ ("Optetrak® HF", Exactech, Gainesville, FL) knee designs. The null hypothesis is that there is no difference in postoperative knee flexion between the Optetrak® PS and Optetrak® HF groups.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is indicated for total knee replacement with a posterior stabilized device.
2. Patient is between the ages of 50 and 80 years old
3. Patient has a Body Mass Index (BMI) < 35.0 using the following method (or comparable method)

   • BMI = Weight (lbs.) ÷ Height (in.)2 x 703
4. Patient is skeletally mature.
5. Patient is willing to participate by complying with pre and postoperative visit requirements, over at least a 1-year period, including completion of studyrequired questionnaires.
6. Patient is willing and able to review and sign a study Informed Consent.

Exclusion Criteria:

1. Patient has a Body Mass Index (BMI) > 35.0 using the following method (or comparable method)

   • BMI = Weight (lbs.) ÷ Height (in.)2 x 703
2. Patient is skeletally mature
3. Patient is willing to participate by complying with pre and postoperative visit requirements, over at least a 1-year period, including completion of study required questionnaires.
4. Patient is willing and able to review and sign a study Informed Consent.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-12 (Estimated); Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
The primary outcome of interest is knee range of motion (ROM), specifically the degree of flexion. | 2 years
  Physician assess range of motion in knee joint

SECONDARY OUTCOMES:
Knee Society Score (KSS) | 2 years
  Validated physician assessed outcome
Hospital for Special Surgery (HSS) Knee Score | 2 years
  Validated physician assessed outcome
Patient Satisfaction | 2 years
  Visual Analog Scale (1-10) where 10 is best.
Implant survivorship | 2 years
  Implant survivorship
Radiographic evaluation | 2 years
  Radiographic analysis
Complications | 2 years
  Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Jason Drenning, Ph.D., Study Director — Exactech; John W. Aldridge, MD, Principal Investigator — Hampton Roads Orthopedics
Locations (1):
- Hampton Roads Orthopedics, Newport News, Virginia, United States